CLINICAL TRIAL: NCT00798018
Title: Effect of Intra-cuff Lidocaine and Tetracaine on Tracheal Tube-induced Emergence Phenomena
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Dr., Department of Anesthesiology, West China Second Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ICLT
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Results first posted 2009-12-18 (Estimated); Last update posted 2009-12-18 (Estimated); Status verified 2009-11

CONDITIONS: Pharyngitis
Keywords: lidocaine; tetracaine; tracheal intubation; pharyngitis
MeSH Terms: conditions — Pharyngitis | interventions — Lidocaine; Tetracaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Air (Placebo Comparator): air was used to inflate the cuff.
  Interventions: Drug: placebo
- Normal Saline (Placebo Comparator): Normal saline was used to inflate the cuff.
  Interventions: Drug: N.S
- lidocaine (Active Comparator): 2% lidocaine was used to inflate the cuff.
  Interventions: Drug: 2% lidocaine
- tetracaine (Experimental): 1% tetracaine was used to inflate the cuff.
  Interventions: Drug: 1% tetracaine

INTERVENTIONS:
Drug: 2% lidocaine — lidocaine: 2%, injected into the cuff to seal the space between the trachea and the tube at minimal volume
  Arms: lidocaine
Drug: placebo — Air injected into the cuff to seal the space between the trachea and the tube at minimal volume
  Arms: Air
Drug: 1% tetracaine — tetracaine: 1%, injected into the cuff to seal the space between the trachea and the tube at minimal volume
  Arms: tetracaine
Drug: N.S — 0.9% Normal saline injected into the cuff to seal the space between the trachea and the tube at minimal volume
  Arms: Normal Saline

SUMMARY:
It has been proven that tracheal tube inflated with lidocaine could decrease the post-intubation sore throat in nitrous oxide anesthesia. In the study, the investigators would like to evaluate the effect of lidocaine inflation in non-nitrous oxide anesthesia and compare the effect of tetracaine, the best mucosal local anesthetics with lidocaine.

DETAILED DESCRIPTION:
The female patients receiving gynecological surgeries were divided into air, saline and 2% lidocaine and 1% tetracaine groups of 25 each using sealed envelope technique. The cuff of the endotracheal tube was inflated by the inflation medium (with the help of intracuff pressure monitoring device) to occlude the leak around the tube by the Minimal Occlusive Volume Technique. This was done by the same anaesthesiologist in all the patients. The cuff volume and pressure were then recorded. The primary outcome of the study was to evaluate the post-intubation sore throat using the visual analogue scale 6h, 24h and 48h after extubation. The secondary outcomes were incidence of complications during emergence of anesthesia and after extubation. Intra-cuff pressure monitoring was done with a pressure monitor, which consisted of the pressure gauge, three-way stopcock whose one end was attached to the pressure monitoring line. Net volume of the inflation medium was noted. Volume of the inflation medium, intra cuff pressure, duration from intubation to extubation and volume of the inflation medium withdrawn from the cuff was noted. Incidence (Yes/No) of tube intolerance, coughing on tube, restlessness, hoarseness, sore throat, breathlessness and laryngospasm were analyzed by the anaesthesiologist who did not know which group the patient belonged to.

ELIGIBILITY:
Inclusion Criteria:

* patients of the age group 18-60 years
* patients belonging to ASA grade I and II undergoing gynecological surgeries in supine position under general anesthesia with controlled ventilation using Poly Vinyl Chloride ETT (same type and make in all patients)

Exclusion Criteria:

* anticipated difficult intubation
* more than one attempt for intubation
* need for naso gastric tube
* episode of coughing and straining
* history of respiratory tract infection and smoking

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2008-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Han Huang, M.D, Principal Investigator — Department of Aensthesiology, West China 2nd Hospital, Sichuan University
Locations (1):
- Department of Anesthesiology, West China Second Hospital, Sichuan University, Chengdu, Sichuan, China

REFERENCES:
- [Background] Estebe JP, Delahaye S, Le Corre P, Dollo G, Le Naoures A, Chevanne F, Ecoffey C. Alkalinization of intra-cuff lidocaine and use of gel lubrication protect against tracheal tube-induced emergence phenomena. Br J Anaesth. 2004 Mar;92(3):361-6. doi: 10.1093/bja/aeh078. PMID 14970135

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started in November 2008 and finished in February 2009, in total 100 patients were enrolled and all of them finished this study.
Groups:
- Air Alone: Only air was injected into the cuff, as the routine practice
- Lidocaine: 2% lidiocaine was used to inflate the cuff
Period: Overall Study
Arm/Group | Air Alone | Normal Saline | Lidocaine | Tetracaine
Started | 25 | 25 | 25 | 25
Completed | 25 | 25 | 25 | 25
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Air Alone | Normal Saline | Lidocaine | Tetracaine | Total
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 25 | 25 | 100
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 39 (8) | 44 (9) | 42 (7) | 41 (10) | 42 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 25 | 25 | 100
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 25 | 25 | 25 | 25 | 100

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale(0-100mm) by the Subject.
Description: visual analogue scale (VAS) was used to evaluate the post-intubation sore throat. The VAS was a well-recongnized standard tool for rating of pain. The VAS measures exactly 100 mm. 0 means no pain and 100 means the worst pain that one can image. Patient marks a point on the line that matches the amount of pain he or she feels.
Time Frame: 6 hours, 12 hours, 24 hours, 48 hours after extubation
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Air Alone | Normal Saline | Lidocaine | Tetracaine
Number analyzed (Participants) | 25 | 25 | 25 | 25
mm
  6h | 51 (37) | 40 (31) | 22 (17) | 9 (8)
  12h | 50 (33) | 38 (19) | 25 (15) | 13 (7)
  24h | 43 (39) | 41 (30) | 20 (18) | 7 (5)
  48h | 45 (36) | 43 (25) | 23 (19) | 9 (4)

ADVERSE EVENTS:
Arm/Group | Air Alone | Normal Saline | Lidocaine | Tetracaine
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes